CLINICAL TRIAL: NCT02925065
Title: Impact of Non-traditional Guitar Group Instruction on Functional Movement and Well-being in Parkinson's Disease Patients
Acronym: PD/Guitar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00091797
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; Non-traditional guitar instruction; Guitar therapy; Upper extremity motor function; Hand dexterity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to early-start or late start guitar groups. Following baseline assessment week, the early-start group will receive twice-weekly non traditional guitar instruction for 6 weeks. The late-start guitar group will receive same intervention after the early-start group complete their 6 week instruction. Study assessments will be conducted during week 7 and week 14. Follow up assessment will be conducted in week 20.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-start guitar instruction group (Experimental): A 6 week twice-weekly non-traditional group guitar instruction will be implemented in addition to usual treatment between weeks 1-6 of the study.
  Interventions: Other: Non-traditional group guitar instruction
- Delayed-start guitar instruction group (Experimental): A 6 week twice-weekly non-traditional group guitar instruction will be implemented in addition to usual treatment between weeks 8-13 of the study.
  Interventions: Other: Non-traditional group guitar instruction

INTERVENTIONS:
Other: Non-traditional group guitar instruction — A 6-week curriculum for non-traditional training in finger-style guitar has been developed with rhythmic and goal oriented upper extremity and finger movements. Guitar group intervention will be implemented at the Towson campus of the Peabody Preparatory. Intervention approaches will include rhythmic digital grip with finger isolation, goal directed rhythmic reach on the fret-board and rhythmic alternating tap-like digit and hand movements on the guitar. Participants will be provided with the instruments in the group setting without expectation of practice at home.

SUMMARY:
This controlled prospective cohort study is designed to assess the feasibility and effect of twice-weekly 60 minute non-traditional guitar classes on PD patient's self-reported and measurable outcomes including upper extremity function, motor findings, quality of life, mood, and cognitive findings. 24-30 individuals with PD will be randomly assigned to an early-start and a late-start guitar instruction group. Prior to conducting a larger study, this study seeks to assess the possibility that participation in an instrumental performance activity in a group setting may improve outcomes in PD patients.

DETAILED DESCRIPTION:
PROBLEM STATEMENT: Engagement in musical activities has been found to improve symptoms in individuals with Parkinson's disease (PD), and physical therapy and music therapy have been demonstrated as viable non-pharmacological intervention methods that improve motor function in these individuals. Therapeutic instrumental music performance has the attributes of physical, rhythmic and social engagement combined with immediate auditory feedback, and has the potential to bring in additional neuro-rehabilitative effects associated with musical engagement into a treatment design. However, until now, much of the research has focused on the rhythmic aspects of music. Few studies have examined how active and complex engagement with music, such as learning to play an instrument, may help PD patients. Finger-style guitar instruction has the potential to improve bilateral dexterity in addition to other gains reported with music-based interventions in patients with PD.

PURPOSE: The purpose of this pilot controlled prospective cohort study is to assess the feasibility and the effects of non-traditional finger-style guitar classes on the quality of life, motor symptoms, upper extremity function, cognition, mood and social participation in individuals with PD.

HYPOTHESIS: The investigators hypothesize that a 6-week bi-weekly finger-style guitar group intervention (12 sessions in total) in addition to usual and routine treatment will be a feasible intervention in patients with Parkinson's Disease (PD), and both immediate and delayed start groups, of PD patients who participate in a twice-weekly non-traditional guitar class training for 6 weeks will have unchanged or improved upper extremity function and dexterity, improved quality of life and mood.

IMPORTANCE: The estimated overall prevalence of PD in the world is 315 per 100,000 individuals overall, and about 2 per 100 individuals 60 years of age or older, with higher estimates for older individuals living in North America, Europe and Australia. PD prevalence in the United States is projected to rise by 77% between 2010 and 2030. Music and rhythm-based interventions are noninvasive, patient-oriented techniques that lack side effects. The guitar is the most popular played instrument in the U.S, and it is the principal instrument of choice for music therapists. It is affordable and portable, with easy access to commercial instruction. Non-traditional engagement in finger-style music making on the guitar may have a broad impact on PD by improving the quality of functional upper extremity movements, decreasing the amplitude of involuntary movements, increasing social and cognitive participation in activities of daily living, and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-89) with idiopathic PD diagnosis according to the United Kingdom (UK) Brain Bank Criteria with bilateral motor symptoms.
* Hoehn and Yahr Stages 1-3.
* MoCA score >24 to screen out patients with dementia.

Exclusion Criteria:

* Prior exposure to guitar training.
* History of prior trauma of the brain or upper extremities.
* Inability to personally consent to study.
* Inability or unwillingness to participate in twice weekly classes for 6 weeks.
* Agitation or hallucinations.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 weeks
  Percentage of study completion will be used to assess feasibility of the intervention along with descriptive statistics. The study will be deemed feasible if 80% of participants complete 10 or more guitar group interventions. The factors that affect probability of attending guitar classes will also be investigated.

SECONDARY OUTCOMES:
Efficacy: Quality of Life | 6 weeks and 12 week follow up
  The Parkinson disease quality of life assessment (PDQ-39) (Peto, Jenkinson & Fitzpatrick, 1998) is a questionnaire that is designed to assess PD specific health related quality of life within the last month in individuals with PD. Dimensions covered include mobility, activities of daily living, emotional well-being, stigma and social support, cognition, communication and bodily support.
Upper extremity motor function | 6 weeks and 12 weeks follow up
  Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Fine manual dexterity | 6 weeks and 12 weeks follow up
  Purdue pegboard test (PPBT) involves timed assembly of small items and assesses fine manual dexterity.
Gross manual dexterity | 6 weeks and 12 weeks follow up
  Box and block test (BBT) involves timed transfer of 2.5cm3 blocks from one container to another and assesses the gross manual dexterity.
Upper extremity activities of daily living function | 6 weeks and 12 weeks follow up
  Quick-Disability of Arm, Shoulder and Hand (Q-DASH) (Gummeson, Ward & Atroshi, 2006) is an 11-item questionnaire that measures the self-reported disability of upper extremity.
Upper extremity finger typing accuracy and speed | 6 weeks and 12 weeks follow up
  Finger typing task: Using index and middle finger to press 2 adjacent standard keyboard keys ('n' and 'm' for the right hand; 'c' and 'v' for the left hand) in alternating fashion as rapidly and accurately as possible in 60 seconds (each hand tested separately).
Cognition | 6 weeks and 12 week follow up
  Montreal Cognitive Assessment (MoCA) (Nasreddine, 2005) is a rapid cognitive screening test that assesses cognitive performance in multiple domains including visuo-spatial and executive functions, naming, memory, attention, language, abstraction, and orientation.
Mood | 6 weeks and 12 week follow up
  Geriatric Depression Scale (GD S-15) (Sheikh & Yesavage, 1986) is a 15 item questionnaire that assesses depression and suicide ideation in elderly individuals.
Social Participation | 6 weeks and 12 weeks follow up
  World Health Organization Disability Assessment Schedule (WHODAS 2.0) Social participation subscale. WHODAS 2.0 is a 36 item disability assessment questionnaire developed by the WHO Classification, Terminology and Standards team to measure health and disability. The social participation subscale (Domain 6) contains 8 items and measures impact of health on social participation.
Group participation | 6 weeks and 12 weeks follow up
  Pittsburg Rehabilitation Participation Scale (PRPS) will be used to monitor participation intensity and quality of the participants in the guitar group intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Serap E Bastepe-Gray, MD, MM, MsOT, Principal Investigator — Johns Hopkins University; Alexander Pantelyat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (Peabody Institute & Department of Neurology), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altenmuller E, Marco-Pallares J, Munte TF, Schneider S. Neural reorganization underlies improvement in stroke-induced motor dysfunction by music-supported therapy. Ann N Y Acad Sci. 2009 Jul;1169:395-405. doi: 10.1111/j.1749-6632.2009.04580.x. PMID 19673814
- [Background] Austin D, Jimison H, Hayes T, Mattek N, Kaye J, Pavel M. Measuring motor speed through typing: a surrogate for the finger tapping test. Behav Res Methods. 2011 Dec;43(4):903-9. doi: 10.3758/s13428-011-0100-1. PMID 21494919
- [Background] Benoit CE, Dalla Bella S, Farrugia N, Obrig H, Mainka S, Kotz SA. Musically cued gait-training improves both perceptual and motor timing in Parkinson's disease. Front Hum Neurosci. 2014 Jul 7;8:494. doi: 10.3389/fnhum.2014.00494. eCollection 2014. PMID 25071522
- [Background] Bloem BR, de Vries NM, Ebersbach G. Nonpharmacological treatments for patients with Parkinson's disease. Mov Disord. 2015 Sep 15;30(11):1504-20. doi: 10.1002/mds.26363. Epub 2015 Aug 14. PMID 26274930
- [Background] de Dreu MJ, van der Wilk AS, Poppe E, Kwakkel G, van Wegen EE. Rehabilitation, exercise therapy and music in patients with Parkinson's disease: a meta-analysis of the effects of music-based movement therapy on walking ability, balance and quality of life. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1:S114-9. doi: 10.1016/S1353-8020(11)70036-0. PMID 22166406
- [Background] Dorsey ER, George BP, Leff B, Willis AW. The coming crisis: obtaining care for the growing burden of neurodegenerative conditions. Neurology. 2013 May 21;80(21):1989-96. doi: 10.1212/WNL.0b013e318293e2ce. Epub 2013 Apr 24. PMID 23616157
- [Background] Francois C, Grau-Sanchez J, Duarte E, Rodriguez-Fornells A. Musical training as an alternative and effective method for neuro-education and neuro-rehabilitation. Front Psychol. 2015 Apr 28;6:475. doi: 10.3389/fpsyg.2015.00475. eCollection 2015. PMID 25972820
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Grau-Sanchez J, Amengual JL, Rojo N, Veciana de Las Heras M, Montero J, Rubio F, Altenmuller E, Munte TF, Rodriguez-Fornells A. Plasticity in the sensorimotor cortex induced by Music-supported therapy in stroke patients: a TMS study. Front Hum Neurosci. 2013 Sep 3;7:494. doi: 10.3389/fnhum.2013.00494. eCollection 2013. PMID 24027507
- [Background] Gummesson C, Ward MM, Atroshi I. The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): validity and reliability based on responses within the full-length DASH. BMC Musculoskelet Disord. 2006 May 18;7:44. doi: 10.1186/1471-2474-7-44. PMID 16709254
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4. doi: 10.1007/pl00007730. PMID 9617716
- [Background] Pohl P, Dizdar N, Hallert E. The Ronnie Gardiner Rhythm and Music Method - a feasibility study in Parkinson's disease. Disabil Rehabil. 2013;35(26):2197-204. doi: 10.3109/09638288.2013.774060. Epub 2013 Mar 12. PMID 23480646
- [Background] Proud EL, Miller KJ, Bilney B, Balachandran S, McGinley JL, Morris ME. Evaluation of measures of upper limb functioning and disability in people with Parkinson disease: a systematic review. Arch Phys Med Rehabil. 2015 Mar;96(3):540-551.e1. doi: 10.1016/j.apmr.2014.09.016. Epub 2014 Oct 7. PMID 25301441
- [Background] Pringsheim T, Jette N, Frolkis A, Steeves TD. The prevalence of Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2014 Nov;29(13):1583-90. doi: 10.1002/mds.25945. Epub 2014 Jun 28. PMID 24976103
- [Background] Raglio A. Music Therapy Interventions in Parkinson's Disease: The State-of-the-Art. Front Neurol. 2015 Aug 31;6:185. doi: 10.3389/fneur.2015.00185. eCollection 2015. No abstract available. PMID 26379619
- [Background] Rochester L, Baker K, Hetherington V, Jones D, Willems AM, Kwakkel G, Van Wegen E, Lim I, Nieuwboer A. Evidence for motor learning in Parkinson's disease: acquisition, automaticity and retention of cued gait performance after training with external rhythmical cues. Brain Res. 2010 Mar 10;1319:103-11. doi: 10.1016/j.brainres.2010.01.001. Epub 2010 Jan 11. PMID 20064492
- [Background] Schneider S, Schonle PW, Altenmuller E, Munte TF. Using musical instruments to improve motor skill recovery following a stroke. J Neurol. 2007 Oct;254(10):1339-46. doi: 10.1007/s00415-006-0523-2. Epub 2007 Jan 27. PMID 17260171
- [Background] Van Vugt FT, Ritter J, Rollnik JD, Altenmuller E. Music-supported motor training after stroke reveals no superiority of synchronization in group therapy. Front Hum Neurosci. 2014 May 20;8:315. doi: 10.3389/fnhum.2014.00315. eCollection 2014. PMID 24904358
- [Background] Hartigan, B. J., & Sarrafian, S. K. (2004). Kinesiology and functional characteristics of upper limb. In D. G. Smith, J. W. Michael, & J. H. Bowker (Eds.), Atlas of amputations and limb deficiencies: surgical, prosthetic, and rehabilitation principles (3rd Edition ed., pp. 101-116). Rosemont, IL: American Academy of Orthopaedic Surgeons.
- [Background] Sheikh J.I., & Yesavage J.A. (1986): Geriatric Depression Scale (GDS): Recent evidence and development of a shorter version. In: Brink TL, editor. Clinical Gerontology: A Guide to Assessment and Intervention. Binghampton,NY: The Haworth Press. 165-173.
- [Background] Richard K Miller and Associates. (2012). The 2012-2013 Leisure Market Research Handbook. Loganville, GA: Richard K. Miller and Associates.